CLINICAL TRIAL: NCT06205030
Title: Efficacy of a Traditional Anti-diabetic Herbal Drug on Glycemic, Inflammatory, and Oxidative Stress Parameters in Patients With Type 2 Diabetes
Brief Title: Efficacy of NOSHINtrial in Diabetic Patients
Acronym: NOSHIN
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kerman Medical University (Other)
Collaborators: Afzalipour Hospital (Other)
Responsible Party: Principal Investigator, Faegheh Bahri, principle investigator, Kerman Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 402000209
Record Dates: First submitted 2023-12-19; First posted 2024-01-12 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance
Keywords: Type 2; Diabetes mellitus; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: All the volunteers who meet the entry criteria were directed to the laboratory so that biochemical tests can be performed on them before taking the drug. Volunteers are asked to take the received medicine three times a day after food. they will be divided into two groups by a person outside the research team, one group will drink herbal syrup and the other group will receive a placebo. A placebo with the same appearance as herbal syrup will drink nectar. On a weekly basis, the researcher will make phone calls with the applicants and, while reminding and recording the amount of herbal syrup consumed by drinking nectar, will also ask about the possible side effects of consuming herbal syrup drinking nectar. Then, at the end of the six week, the patient was asked to visit the clinic for a final evaluation.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Anti-diabetic herbal and placebo syrups with the same color, shape, and box but different codes in two groups A and B are employed. After enrollment, each patient is allocated a code. Patients, researchers, and physicians who collect information in this study, assess outcomes, and analyze data for the study are blinded to the assigned treatment (anti-diabetic herbal or placebo) so that all patients are evaluated using their specific assigned code and treatment groups A or B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NOSHIN SHAHD drug (Active Comparator): All the volunteers directed to the laboratory so that biochemical tests can be performed on them before taking the drug. Volunteers are asked to take the received NOSHIN SHAHD drug 20 ml three times per day after food. at the end of the six week. then, the sample collection will be done to review all the tests of the end stage of receiving the drug.
  Interventions: Drug: anti-diabetic herbal drug
- placebo (Placebo Comparator): The placebo with the same appearance as the herbal syrup will be drinking nectar. All the volunteers directed to the laboratory so that biochemical tests can be performed on them before taking the drug. Volunteers are asked to take the received placebo 20 ml three times per day after food. at the end of the six week. then, the sample collection will be done to review all the tests of the end stage of receiving the drug.
  Interventions: Drug: anti-diabetic herbal drug

INTERVENTIONS:
Drug: anti-diabetic herbal drug — All the volunteers directed to the laboratory so that biochemical tests can be performed on them before taking the drug. Volunteers are asked to take the received NOSHIN SHAHD drug 20 ml three times per day after food. at the end of the six week. then, the sample collection will be done to review all the tests of the end stage of receiving the drug.
  Other Names: NOSHIN SHAHD drug

SUMMARY:
The goal of this [Efficacy of a traditional anti-diabetic herbal drug with on glycemic, inflammatory, and oxidative stress parameters] is [investigate the level of HOMA-estimated insulin resistance as the primary outcome before and after 40 days in intervention and placebo groups] in [patients with type 2 diabetes]. The secondary outcomes of this study are the assessment of oxidative stress, inflammation biomarkers, other glycemic indices, hematopoietic status and lipid profile between the two groups before and after the intervention. also The food frequency questionnaire (FFQ) and the physical activity questionnaire (FAQ) are used to evaluate the effect of potential confounding factors. This study has the code of ethics IR.KMU.REC.1402.291 from Kerman University of Medical Sciences and this drug has the number 12/14484 from Iran Food and Drug Administration (IFDA).

DETAILED DESCRIPTION:
All the volunteers (Diabetic men and women with HbA1c more than 6.5 from the age of 20 to 65 years who usually use their standard medicine) who meet the entry criteria were directed to the laboratory and imaging center so that biochemical tests can be performed on them before taking the drug. Volunteers are asked to take the received medicine three times a day after food. It is worth mentioning that the patients will be divided into two groups by a person outside the research team, one group will drink herbal syrup and the other group will receive a placebo. A placebo with the same appearance as herbal syrup will drink nectar. On a weekly basis, the researcher will make phone calls with the applicants and, while reminding and recording the amount of herbal syrup consumed by drinking nectar, will also ask about the possible side effects of consuming herbal syrup drinking nectar. Then, at the end of the six week, the patient was asked to visit the clinic for a final evaluation. In this stage, the patient is asked about possible side effects, and the last stage of sample collection will be done to review all the tests of the next stage of receiving the drug (biochemical tests). Return at the end of week 6. The sample size in this study is 70 people.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 65 years
2. HbA1c more than 6.5
3. Consistency of diet and exercise program
4. Body mass index less than 35
5. Not receiving insulin
6. The patient should take standard medicine except insulin

Exclusion Criteria:

1. Performing CABG surgery, occurrence of ASC, heart and brain stroke, pulmonary embolism, deep vein thrombosis or TIA in the last 1 year.
2. Taking anti-inflammatory drugs such as aspirin with an anti-inflammatory dose, antioxidant supplements, vitamins and omega-3 capsules (<1 g/day), and immunosuppressive drugs in the last three months.
3. Presence of cancer, liver and thyroid diseases.
4. pregnancy
5. Smoking and alcohol consumption

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-26 (Estimated); Primary Completion 2027-07-16 (Estimated); Study Completion 2027-08-16 (Estimated)

PRIMARY OUTCOMES:
HOMA-estimated insulin resistance | 40 days
  To investigate the effect of the anti-diabetic herbal drug on changes in HOMA-IR in patients with T2DM

SECONDARY OUTCOMES:
plasma MDA | 40 days
  Investigating the changes in plasma Malondialdehyde level as an oxidative stress factor
plasma protein carbonyl | 40 days
  Investigating the changes in plasma protein carbonyl level as an oxidative stress factor
plasma TAC | 40 days
  Investigating the changes in plasma total antioxidant capacity as an oxidative stress factor
plasma SOD enzyme activity | 40 days
  Investigating the changes in plasma SOD enzyme activity as an oxidative stress factor
plasma catalase enzyme activity | 40 days
  Investigating the changes in plasma catalase enzyme activity as an oxidative stress factor
plasma reduced glutathione | 40 days
  Investigating the changes in plasma reduced glutathione levels as an oxidative stress factor
ROS in PBMCs | 40 days
  Investigating the changes in ROS level in PBMCs as an oxidative stress factor
FBS | 40 days
  Investigating the changes in fasting blood glucose as a glycemic status
fasting blood Insulin | 40 days
  Investigating the changes in fasting blood Insulin as a glycemic status
HbA1c | 40 days
  Investigating the changes in HbA1c level as a glycemic status
Inflammatory biomarkers | 40 days
  Investigating the changes in plasma TNF-α, IL-6, IL-1β, and hs-CRP levels

OTHER OUTCOMES:
WBC count | 40 days
  Investigating the changes in White blood cell counts as hematopoietic status
RBC count | 40 days
  Investigating the changes in Red blood cell counts as a hematopoietic status
Hemoglobin | 40 days
  Investigating the changes in hemoglobin level as a hematopoietic status
Hematocrit | 40 days
  Investigating the changes in hematocrit level as a hematopoietic status
blood MCV | 40 days
  Investigating the changes in amount of MCV level as a hematopoietic status
blood MCH | 40 days
  Investigating the changes in amount of MCH level as a hematopoietic status
blood MCHC | 40 days
  Investigating the changes in amount of MCHC level as a hematopoietic status
serum Urea | 40 days
  Investigating the changes in serum Urea level as a biochemistry factor
serum Uric acid | 40 days
  Investigating the changes in serum Uric acid level as a biochemistry factor
serum Creatinine | 40 days
  Investigating the changes in serum Creatinine level as a biochemistry factor
BUN | 40 days
  Investigating the changes in Blood urea nitrogen level as a biochemistry factor
Total protein | 40 days
  Investigating the changes in total protein level as a biochemistry factor
Albumin | 40 days
  Investigating the changes in Albumin level as a biochemistry factor
ALT | 40 days
  Investigating the changes in Alanine transaminase level as a biochemistry factor
AST | 40 days
  Investigating the changes in Aspartate Aminotransferase level as a biochemistry factor
lipid profile | 40 days
  Investigating the changes in serum triglyceride, LDL cholesterol, HDL cholesterol, and Total cholesterol levels

CONTACTS AND LOCATIONS:
Locations (1):
- Kerman University of Medical Sciences, Kerman, Iran

IPD SHARING:
Plan to Share IPD: Yes
A part of the data such as the information related to the main outcome or the like can be shared. Access to study documentation after results are published and It will be available for researchers working in academic and scientific institutions, and also people who are working in the industry can apply for them for secondary studies. The request sent will be reviewed by the members of the center. If the members agree, they will be notified.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Access to study documentation after results are published.
Access Criteria: It will be available for researchers working in academic and scientific institutions, and also people who are working in the industry can apply for them for secondary studies.
URL: https://isid.research.ac.ir/Hossein_Pourghadamyari